CLINICAL TRIAL: NCT02785900
Title: A Randomized, Double-blind Phase 3 Study of Vadastuximab Talirine (SGN-CD33A) Versus Placebo in Combination With Azacitidine or Decitabine in the Treatment of Older Patients With Newly Diagnosed Acute Myeloid Leukemia (AML)
Brief Title: Vadastuximab Talirine (SGN-CD33A; 33A) Combined With Azacitidine or Decitabine in Older Patients With Newly Diagnosed Acute Myeloid Leukemia
Acronym: CASCADE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to safety; specifically a higher rate of deaths, including fatal infections, in the SGN33A arm versus the control arm
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SGN33A-005; 2015-003482-28 (EudraCT Number)
Record Dates: First submitted 2016-05-25; First posted 2016-05-30 (Estimated); Results first posted 2018-12-12 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-11

CONDITIONS: Acute Myeloid Leukemia
Keywords: Antibodies, monoclonal; Antibody drug conjugate; Antigens, cluster of differentiation 33 (CD33); Drug therapy; Immunotherapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — vadastuximab talirine; Azacitidine; Decitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 33A + HMA (Experimental): 33A plus azacitidine or decitabine
  Interventions: Drug: 33A; Drug: azacitidine; Drug: decitabine
- placebo + HMA (Active Comparator): placebo plus azacitidine or decitabine
  Interventions: Drug: placebo; Drug: azacitidine; Drug: decitabine

INTERVENTIONS:
Drug: 33A — 33A, 10 mcg/kg, every 4 weeks via intravenous (IV) push
  Other Names: vadastuximab talirine, SGN-CD33A
  Arms: 33A + HMA
Drug: placebo — Volume equivalent to 10 mcg/kg, every 4 weeks via IV push
  Arms: placebo + HMA
Drug: azacitidine — 75 mg/m2 given subcutaneously (SC) or IV x 7 days, every 4 weeks
Drug: decitabine — 20 mg/m2 given IV x 5 days, every 4 weeks

SUMMARY:
The purpose of this study in AML patients is to test whether vadastuximab talirine (SGN-CD33A; 33A) combined with either azacitidine or decitabine improves remission rates and extends overall survival as compared to placebo combined with either azacitidine or decitabine.

DETAILED DESCRIPTION:
Hypomethylating agents (HMAs), such as decitabine or azacitidine, are considered a standard treatment for older patients with AML. The primary goals of this study are to test whether patients treated with an HMA (either decitabine or azacitidine) in combination with 33A will have better anti-tumor activity and/or survive longer than patients treated with an HMA in combination with placebo.

Patients who meet eligibility criteria will be randomly assigned to one of two treatment groups: 1) 33A plus HMA (Experimental Arm); or 2) placebo plus HMA (Comparator Arm). In addition to evaluating survival and remission rates, the minimal residual disease (MRD)-negative remission rate, duration of remission, event free- and leukemia-free survival, and safety and tolerability will be compared between arms.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, previously untreated, cytologically/histologically confirmed de novo or secondary AML according to World Health Organization (WHO) classification (except for acute promyelocytic leukemia (APL))
* Intermediate or adverse cytogenetic risk
* Eligible for therapy with either decitabine or azacitidine
* Acceptable hematologic and organ function

Exclusion Criteria:

* AML associated with favorable risk karyotypes including inv(16), t(8;21), t(16;16), or t(15;17)
* Patients who are candidates for allogeneic stem cell transplant at the time of enrollment
* Patients with a history of one of the following myeloproliferative neoplasms: essential thrombocythemia, polycythemia vera, and primary myelofibrosis
* Received prior treatment with HMA or chemotherapy for antecedent myelodysplastic syndrome (MDS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2016-05; Primary Completion 2017-10-03 (Actual); Study Completion 2017-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phoenix Ho, MD, Study Director — Seagen Inc.
Locations (128):
- United States (40):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope National Medical Center, Duarte, California
  - Pacific Hematology Oncology Associates, San Francisco, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Florida Cancer Specialists - South Region, Fort Myers, Florida
  - Shands Cancer Center / University of Florida, Gainesville, Florida
  - Memorial Cancer Institute, Miami, Florida
  - Florida Center for Cellular Therapy / Blood and Marrow Transplant Center, Orlando, Florida
  - Florida Cancer Specialists - North Region, St. Petersburg, Florida
  - Northside Hospital, Atlanta, Georgia
  - OnCare Hawaii, Honolulu, Hawaii
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Kansas Cancer Center, Westwood, Kansas
  - Norton Cancer Institute, Louisville, Kentucky
  - LSU Health Sciences Center / Feist Weiller Cancer Center, Shreveport, Louisiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - James P. Wilmot Cancer Center / University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Providence Portland Medical Center, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina/Hollings Cancer Center, Charleston, South Carolina
  - Saint Francis Hospital / Bon Secours, Greenville, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center / University of Texas, Houston, Texas
  - Brooke Army Medical Center, San Antonio, Texas
  - Texas Oncology - San Antonio Medical Center, San Antonio, Texas
  - Intermountain Blood and Marrow Transplant/Acute Leukemia Program, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - Swedish Cancer Institute, Seattle, Washington
- Australia (5):
  - Royal Adelaide Hospital, Adelaide
  - Monash Medical Centre, Clayton
  - St George Hospital, Kogarah
  - Royal Perth Hospital, Perth
  - Sunshine Hospital, St Albans
- Austria (2):
  - LKH Salzburg, Universitatsklinikum der PMU, Salzburg
  - Klinikum Wels-Grieskirchen GmbH, Wels
- Belgium (7):
  - Ziekenhuis Netwerk Antwerpen Campus Stuivenberg, Antwerp
  - Az Sint-Jane Brugge - Oostende Av - Campus Sint-Jan, Bruges
  - Institut Jules Bordet, Brussels
  - Cliniques Universitaires Saint Luc, Brussels
  - Centre Hospitalier Universitaire Sart Tilman Liege, Liège
  - AZ Delta - Campus Wilgenstraat, Roeselare
  - Cliniques Universitaires UCL de Mont-Goddine, Yvoir
- Czechia (4):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove-oddeleni klinicke hematologie, Hradec Králové
  - Fakultni Nemocnice Ostrava, Ostrava - Poruba
  - Ustav hematologie a krevni transfuze, Prague
- France (15):
  - CHU Amiens Picardie - Site Sud, Amiens
  - Center Hospitalier Universitaire d' Angers, Angers
  - Centre Hospitalier Victor Dupouy d'Argenteuil, Argenteuil
  - Centre Hospitalier Universitaire Hopital Avicenne, Bobigny
  - Hopital d'Instruction des Armees - Percy, Clamart
  - CHRU de Lille, Lille
  - Centre Hospitalier Universitaire (CHU) De Limoges - Hopital Dupuytren, Limoges
  - Hopital Emile Muller, Mulhouse
  - Centre Hospitalier Universitaire Nantes-Hotel Dieu, Nantes
  - CHU de Nice - Hopital l'Archet, Nice
  - Hopital Saint-Louis / Service d'Hematologie, Paris
  - CHU Bordeaux Hopital Haut-Levaque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Centre Hospitalier Universitaire de Rennes, Hopital Pontchaillou, Rennes
- Germany (5):
  - Stadtisches Klinikum Braunschweig gGmbH, Braunschweig
  - Universitatsklinikum Koln, Cologne
  - Marien Hospital Dusseldorf GmbH, Düsseldorf
  - Universitatsklinik Freiburg, Freiburg im Breisgau
  - Universitatsklinikum Schleswig-Holstein, Kiel
- Hungary (5):
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem Orvos Ã©s Egeszsegtudomanyi Centrum, III. sz. Belgyogyaszati Klinika, Debrecen
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár
  - Bacs-Kiskun Megyei Korhaz Szegedi Tudomanyegyetem Altalanos Orvostudomanyi Kar Oktato Korhaza, Kecskemét
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikat Kozpont, Szeged
- Israel (8):
  - Barzilai Medical Center, Ashkelon
  - Soroka Medical Center, Dept. of Oncology, Beersheba
  - Carmel Medical Center, Haifa
  - Edith Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (5):
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Azienda Ospedaliero-Univesitaria San Luigi Gonzaga, Orbassano
  - Azienda Ospedaliera Ospedali Riuniti Marche Nord, Pesaro
  - Università degli Studi di Roma "La Sapienza, Policlinico Umberto I, Roma
- Centre Hospitalier Luxembourg - CHL Centre, Luxembourg, Luxembourg
- Poland (2):
  - SPZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - Samodzielny Publiczny Centralny Szpital Kliniczny, Warsaw
- South Korea (10):
  - Keimyung University Dongsan Medical Center, Daegu
  - Yeungnam University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hwasun Hospital, Hwasun
  - Chonbuk National University Hospital, Jeonju
  - Seoul National University Hospital, Jongno-gu
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Seoul Saint Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (9):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital de la Santa Creu i Sant Paul, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Universitario de Girona Doctor Josep Trueta, Girona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitaro de Salamanca, Salamanca
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Taiwan (4):
  - Changhua Christian Hospital, Changhua
  - National Cheng-Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (6):
  - County Durham and Darlington NHS Foundation Trust, Darlington
  - Imperial College Healthcare NHS Trust, London
  - North West London Hospitals NHS Trust, Middlesex
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - University Hospitals of North Midlands NHS Trust, Stoke-on-Trent

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 33A + HMA | Placebo + HMA
Started | 117 | 123
Completed | 0 | 0
Not Completed | 117 | 123
Not completed — Study Termination by Sponsor | 64 | 81
Not completed — Death | 46 | 32
Not completed — Withdrawal by Subject | 4 | 8
Not completed — Physician Decision | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 33A + HMA | Placebo + HMA | Total
Number analyzed (Participants) | 117 | 123 | 240
Age, Continuous [Median (Full Range); unit: years] | 75.0 [62 to 91] | 75.0 [52 to 91] | 75.0 [52 to 91]
Age, Customized [Count of Participants; unit: Participants]
  Age Group: >65 years | 3 | 3 | 6
  Age Group: 65 - 74 years | 55 | 55 | 110
  Age Group: 75 - 79 years | 33 | 41 | 74
  Age Group: >= 80 years | 26 | 24 | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 67 | 136
  Male | 48 | 56 | 104
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 98 | 111 | 209
  Unknown or Not Reported | 16 | 10 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian | 12 | 16 | 28
  Race: Black or African American | 3 | 1 | 4
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: White | 85 | 94 | 179
  Race: Other | 2 | 1 | 3
  Race: Not Reportable | 13 | 10 | 23
  Race: Unknown | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Hungary | 5 | 6 | 11
  United States | 49 | 45 | 94
  Czechia | 3 | 6 | 9
  United Kingdom | 5 | 3 | 8
  Spain | 5 | 6 | 11
  South Korea | 6 | 7 | 13
  Austria | 3 | 0 | 3
  Belgium | 4 | 8 | 12
  Taiwan | 5 | 5 | 10
  Italy | 2 | 3 | 5
  Israel | 5 | 7 | 12
  France | 13 | 10 | 23
  Australia | 10 | 11 | 21
  Germany | 2 | 6 | 8
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — 0=Normal activity; 1=Symptoms but ambulatory; 2=In bed less than 50% of the time; 3= In bed more than 50% of the time; 4=100% bedridden; 5=Dead
  Participants
    Grade 0: Normal activity | 23 | 23 | 46
    Grade 1: Symptoms but ambulatory | 78 | 80 | 158
    Grade 2: In bed less than 50% of the time | 16 | 20 | 36

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Time from randomization to death due to any cause
Time Frame: Up to 1.5 years
Population: Intent-to-treat analysis set
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | 33A + HMA | Placebo + HMA
Number analyzed (Participants) | 117 | 123
months | 5.1 [2.3 to 9.9] | NA [4.0 to NA] — Insufficient number of participants with events

2. Primary Outcome: Composite Complete Remission (CRc) Rate
Description: Number of patients who achieved complete remission (CR) or complete remission with incomplete blood count recovery (CRi) according to the modified response criteria for acute myeloid leukemia (AML) per Cheson 2003.
Time Frame: Up to 1.5 years
Population: Intent-to-treat analysis set
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | 33A + HMA | Placebo + HMA
Number analyzed (Participants) | 117 | 123
participants | 30 [18 to 34.5] | 26 [14.3 to 29.4]

3. Secondary Outcome: Minimal Residual Disease (MRD)-Negative Composite Complete Remission Rate
Description: Number of patients who achieve both remission (CR or CRi) and MRD-negative status
Time Frame: Up to 1.5 years
Population: Intent-to-treat analysis set
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | 33A + HMA | Placebo + HMA
Number analyzed (Participants) | 117 | 123
participants
  MRD-negative CRc rate | 18 [9.4 to 23.2] | 10 [4 to 14.4]
  MRD-negative CR rate | 8 [3 to 13] | 5 [1.3 to 9.2]
  MRD-negative CRi rate | 10 [4.2 to 15.2] | 5 [1.3 to 9.2]

4. Secondary Outcome: Duration of Remission
Description: Duration of remission is calculated from the first documentation of CR or CRi to the first documentation of disease relapse or death, whichever comes first. Patients who are in remission at the time of analysis cutoff are censored at the date of last response assessment. Patients who started another anticancer therapy before relapse or death are censored at the date of last response assessment prior to start of new therapy.
Time Frame: Up to approximately 9.5 months
Population: Patients who achieved complete remission (CR) or CR with incomplete hematologic recovery (CRi).
Measure: Median (Full Range); unit: months
Arm/Group | 33A + HMA | Placebo + HMA
Number analyzed (Participants) | 30 | 26
months | 5.1 [0.03 to 6.21] | 7.5 [0.03 to 9.49]

5. Secondary Outcome: Event-free Survival
Description: Event-free survival is calculated from the time of randomization to the first documentation of progression, relapse, or death, whichever comes first. Patients who do not have event (progression, relapse, or death) prior to analysis cutoff date are censored at the date of last response assessment. Patients who started another anticancer therapy before progression, relapse, or death are censored at the date of last response assessment prior to the start of new therapy. Patients who do not have response assessment post-baseline are censored at the date of randomization.
Time Frame: Up to approximately 11.24 months
Population: Intent-to-treat analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 33A + HMA | Placebo + HMA
Number analyzed (Participants) | 117 | 123
months | 4.2 [3.5 to 5.1] | 6.7 [4.5 to 9.5]

6. Secondary Outcome: Leukemia-free Survival
Description: Leukemia-free survival is calculated from the first documentation of blast clearance (CR, CRi, mLFS) to the first documentation of disease relapse or death, whichever comes first. Patients who are in remission at the time of analysis cutoff are censored at the date of last response assessment. Patients who started another anticancer therapy before relapse or death are censored at the date of last response assessment prior to start of new therapy.
Time Frame: Up to approximately 9.49 months
Population: Patients who achieved CR/CRi
Measure: Median (Full Range); unit: months
Arm/Group | 33A + HMA | Placebo + HMA
Number analyzed (Participants) | 30 | 26
months | 5.1 [0.03 to 8.31] | 7.5 [0.03 to 9.49]

7. Secondary Outcome: Type, Incidence, Severity, Seriousness, and Relatedness of Adverse Events
Description: Treatment-emergent adverse events (TEAEs) are presented and defined as newly occurring (not present at baseline) or worsening after first dose of investigational product. SAE = serious adverse event. "Study treatment" in this data set refers to blinded study treatment.
Time Frame: Up to 1.5 years
Population: Safety analysis set: 7 patients randomized to the HMA+33A received only HMA and are included in the HMA+Placebo safety set. 1 patient randomized to the HMA+placebo arm received 33A+HMA treatment. 1 patient in the HMA+placebo arm did not receive any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | 33A + HMA | Placebo + HMA
Number analyzed (Participants) | 111 | 128
Participants
  Patient with any TEAE | 111 | 125
  Patients with any AE related to study treatment | 83 | 59
  Patients with any SAE | 92 | 89
  Patients with any SAE related to study treatment | 51 | 20
  Patients with Grade 3 or Higher AE | 103 | 112

8. Secondary Outcome: Incidence of Grade 3 or Higher Laboratory Abnormalities
Description: Participants who experienced a laboratory grade increase to Grade 3 or higher (per National Cancer Institute's Common Terminology Criteria for Adverse Events [NCI CTCAE], v4.03)
Time Frame: Up to 1.5 years
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | 33A + HMA | Placebo + HMA
Number analyzed (Participants) | 111 | 128
Participants
  Alanine Aminotransferase (IU/L) - High | 0 | 2
  Albumin (g/dL) - Low | 2 | 4
  Alkaline Phosphatase (IU/L) - High | 0 | 2
  Amylase (IU/L) - High | 1 | 0
  Aspartate Aminotransferase (IU/L) - High | 1 | 2
  Bilirubin (mg/dL) - High | 1 | 1
  Calcium (mg/dL) - Low | 8 | 3
  Creatinine (mg/dL) - High | 0 | 1
  Glucose (mg/dL) - High | 12 | 9
  Magnesium (mg/dL) - High | 2 | 0
  Phosphate (mg/dL) - Low | 17 | 9
  Potassium (mEq/L) - High | 1 | 0
  Potassium (mEq/L) - Low | 5 | 14
  Sodium (mEq/L) - Low | 13 | 12
  Triacylglycerol Lipase (IU/L) - High | 10 | 4
  Urate (mg/dL) - High | 4 | 7
  Hemoglobin (g/dL) - Low | 59 | 66
  Leukocytes (x10^3/uL) - High | 0 | 3
  Leukocytes (x10^3/uL) - Low | 86 | 70
  Lymphocytes (x10^3/uL) - High | 1 | 4
  Lymphocytes (x10^3/uL) - Low | 51 | 29
  Neutrophils (x10^3/uL) - Low | 63 | 43
  Platelets (x10^3/uL) - Low | 77 | 75

9. Secondary Outcome: Time to Complete Remission
Description: Time to CR or CRi is the time from randomization to the first documentation of CR/CRi
Time Frame: Up to 1.5 years
Population: Intent-to-Treat Analysis Set - Patients who Achieved CR/CRi.
Measure: Median (Full Range); unit: weeks
Arm/Group | 33A + HMA | Placebo + HMA
Number analyzed (Participants) | 30 | 26
weeks | 9.3 [5 to 22] | 9.4 [7 to 26]

10. Secondary Outcome: Mortality Rates at Day 30 and Day 60
Description: 30- and 60-day survival from date of randomization. Estimated using Kaplan-Meier method.
Time Frame: Up to 60 days
Population: Intent-to-Treat Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 33A + HMA | Placebo + HMA
Number analyzed (Participants) | 117 | 123
percentage of participants
  30-day Mortality Rate | 11 [7 to 18] | 6 [3 to 12]
  60-day Mortality Rate | 23 [16 to 32] | 13 [8 to 20]

ADVERSE EVENTS:
Time Frame: Up to 13 months
Description: Treatment-emergent adverse events: a newly occurring or worsening adverse event after the first dose of study drug. Safety Analysis Set: 7 patients randomized to the HMA+33A received only HMA and are included in the HMA+Placebo safety set. 1 patient randomized to the HMA+placebo arm received 33A+HMA treatment. 1 patient in the HMA+placebo arm did not receive any study treatment.
Arm/Group | 33A + HMA | Placebo + HMA
All-Cause Mortality (participants affected / at risk) | 43/111 | 34/128
Serious Adverse Events (participants affected / at risk) | 92/111 | 89/128
Other Adverse Events (participants affected / at risk) | 105/111 | 123/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 33A + HMA (N=111) | Placebo + HMA (N=128)
Pneumonia (Infections and infestations) | 22 (24) | 15 (16)
Sepsis (Infections and infestations) | 14 (15) | 7 (10)
Cellulitis (Infections and infestations) | 6 (6) | 8 (8)
Lung infection (Infections and infestations) | 9 (10) | 3 (3)
Septic shock (Infections and infestations) | 6 (6) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 4 (4)
Diverticulitis (Infections and infestations) | 2 (2) | 3 (3)
Bronchitis (Infections and infestations) | 1 (1) | 3 (3)
Bacteraemia (Infections and infestations) | 2 (2) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 3 (3) | 0 (0)
Staphylococcal infection (Infections and infestations) | 2 (2) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 1 (1)
Device related infection (Infections and infestations) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 2 (2) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 2 (2) | 0 (0)
Acinetobacter bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1)
Catheter site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pilonidal cyst (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (1)
Sialoadenitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (2) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 39 (55) | 31 (39)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (7) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 5 (6) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 5 (6) | 0 (0)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 2 (3) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 8 (8) | 8 (8)
General physical health deterioration (General disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 0 (0) | 2 (2)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 2 (2) | 0 (0)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Extravasation (General disorders) | 0 (0) | 1 (1)
Facial pain (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (4)
Neutropenic colitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Palatal oedema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 2 (5)
Cardiac failure (Cardiac disorders) | 2 (2) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Embolism (Vascular disorders) | 2 (2) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Blood culture positive (Investigations) | 1 (1) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
General physical condition abnormal (Investigations) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 4 (4)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Facial paresis (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Serotonin syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Radiation proctitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Vasculitic rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Blood product transfusion dependent (Social circumstances) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 33A + HMA (N=111) | Placebo + HMA (N=128)
Constipation (Gastrointestinal disorders) | 39 (48) | 54 (64)
Nausea (Gastrointestinal disorders) | 37 (49) | 45 (56)
Diarrhoea (Gastrointestinal disorders) | 34 (47) | 34 (52)
Vomiting (Gastrointestinal disorders) | 15 (25) | 31 (41)
Abdominal pain (Gastrointestinal disorders) | 11 (13) | 12 (15)
Mouth ulceration (Gastrointestinal disorders) | 7 (7) | 9 (9)
Stomatitis (Gastrointestinal disorders) | 8 (10) | 6 (7)
Dyspepsia (Gastrointestinal disorders) | 10 (10) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 4 (5) | 7 (7)
Anaemia (Blood and lymphatic system disorders) | 49 (78) | 59 (105)
Thrombocytopenia (Blood and lymphatic system disorders) | 39 (73) | 47 (67)
Neutropenia (Blood and lymphatic system disorders) | 19 (35) | 24 (34)
Febrile neutropenia (Blood and lymphatic system disorders) | 25 (29) | 12 (18)
Leukopenia (Blood and lymphatic system disorders) | 13 (23) | 8 (9)
Oedema peripheral (General disorders) | 33 (38) | 23 (28)
Fatigue (General disorders) | 25 (27) | 24 (25)
Pyrexia (General disorders) | 25 (38) | 18 (31)
Asthenia (General disorders) | 13 (16) | 14 (14)
Injection site erythema (General disorders) | 11 (18) | 4 (6)
Chills (General disorders) | 8 (9) | 4 (5)
Localised oedema (General disorders) | 6 (11) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 28 (43) | 30 (36)
Decreased appetite (Metabolism and nutrition disorders) | 29 (36) | 28 (29)
Hypomagnesaemia (Metabolism and nutrition disorders) | 11 (17) | 13 (16)
Hyponatraemia (Metabolism and nutrition disorders) | 10 (12) | 13 (22)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 9 (10) | 10 (10)
Hypocalcaemia (Metabolism and nutrition disorders) | 10 (11) | 8 (8)
Hypophosphataemia (Metabolism and nutrition disorders) | 8 (10) | 9 (9)
Fluid overload (Metabolism and nutrition disorders) | 3 (3) | 7 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 (20) | 28 (31)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (22) | 20 (25)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 21 (32) | 11 (12)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 12 (15) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 6 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (5)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3)
Weight decreased (Investigations) | 15 (17) | 17 (17)
Platelet count decreased (Investigations) | 12 (19) | 10 (12)
Blood creatinine increased (Investigations) | 9 (10) | 7 (9)
Neutrophil count decreased (Investigations) | 6 (8) | 8 (13)
White blood cell count decreased (Investigations) | 6 (8) | 5 (10)
Blood bilirubin increased (Investigations) | 6 (6) | 1 (1)
Cellulitis (Infections and infestations) | 10 (11) | 10 (10)
Oral candidiasis (Infections and infestations) | 6 (7) | 9 (10)
Pneumonia (Infections and infestations) | 10 (11) | 3 (3)
Oral herpes (Infections and infestations) | 2 (2) | 10 (12)
Urinary tract infection (Infections and infestations) | 4 (4) | 8 (9)
Rash (Skin and subcutaneous tissue disorders) | 11 (15) | 15 (19)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (8) | 13 (13)
Erythema (Skin and subcutaneous tissue disorders) | 3 (4) | 8 (10)
Purpura (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2)
Insomnia (Psychiatric disorders) | 21 (22) | 12 (13)
Confusional state (Psychiatric disorders) | 7 (9) | 7 (7)
Anxiety (Psychiatric disorders) | 8 (8) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (10) | 10 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 9 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (12) | 6 (6)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3)
Hypotension (Vascular disorders) | 12 (12) | 9 (11)
Haematoma (Vascular disorders) | 9 (11) | 9 (12)
Hypertension (Vascular disorders) | 7 (7) | 3 (3)
Dizziness (Nervous system disorders) | 6 (6) | 17 (18)
Headache (Nervous system disorders) | 5 (7) | 17 (18)
Dysgeusia (Nervous system disorders) | 7 (7) | 5 (5)
Contusion (Injury, poisoning and procedural complications) | 11 (14) | 7 (11)
Fall (Injury, poisoning and procedural complications) | 10 (13) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 8 (8) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 7 (7) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 6 (6) | 6 (8)
Urinary retention (Renal and urinary disorders) | 6 (6) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 6 (8) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-12-04): https://cdn.clinicaltrials.gov/large-docs/00/NCT02785900/SAP_000.pdf
  • Study Protocol (2017-03-27): https://cdn.clinicaltrials.gov/large-docs/00/NCT02785900/Prot_001.pdf